CLINICAL TRIAL: NCT03024528
Title: Validation of the Polish Version of CPOT (Critical Care Pain Observation Tool) to Assess Pain Intensity in Adult, Intubated ICU Patients, POL-CPOT.
Brief Title: Validation of the Polish Version of CPOT
Acronym: POL-CPOT
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Kotfis, MD, PhD, DESA, Pomeranian Medical University Szczecin
Other Study IDs: POL-CPOT
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Pain; ICU Delirium
Keywords: Pain; CPOT; ICU Delirium; Critical Care Pain Observation Tool; NRS; Behaviour; Critical care; Intensive Care
MeSH Terms: conditions — Pain; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CAM-ICU (+): Delirious patients.
  Interventions: Behavioral: CPOT assessment
- CAM-ICU (-): Non-delirious patients
  Interventions: Behavioral: CPOT assessment

INTERVENTIONS:
Behavioral: CPOT assessment — Polish version of Critical care pain observation tool validation.
  Other Names: Pain assessment in non-verbal patients

SUMMARY:
Pain experienced by critically ill patients is a major problem affecting nearly 50% of the patients. Assessing pain in critically ill patients is a challenge even in an intensive care unit (ICU) with a minimal opioid-based sedation protocol. In patients who are unable to self-report pain, behavioural scales are used, such as CPOT - Critical Care Pain Observation Tool.

Aim: The aim of this study was to validate the Polish version of a behavioural pain assessment method - CPOT in an ICU with a minimal sedation protocol (opioid-based) versus self-report pain using Numeric rating scale (NRS) in both delirious and non-delirious patients (assessed using Confusion Assessment Method for ICU, CAM-ICU).

Method: A prospective observational cohort study will include 70 patients. The patients will be observed during a non-nociceptive procedure (wash of an arm) and a nociceptive procedure (turning). Patients will be observed 5 minutes before, during, and 15 min after the two interventions (six assessments). Each CPOT assessment will be carried out by two observers blinded to each other. To validate the Polish CPOT translation calculations of interrater reliability, criterion validity and discriminant validity will be performed.

DETAILED DESCRIPTION:
Critically ill patients frequently suffer from pain during their stay in the intensive care unit, as nearly 30% of those patients experience pain at rest and up to 50% experience pain during nursing procedures. Pain experienced by critically ill patients falls into four categories that coexist and overlap: pre-existing chronic pain, acute illness-related pain, continuous ICU treatment-related pain or discomfort and intermittent procedural pain. Moreover, acute pain experienced in the ICU may become a chronic problem after discharge from the unit, as a lifelong ICU footprint. Everyday nursing procedures and interventions (i.e. positioning, mouth and trachea suctioning, wound care, catheter removal or placement, cannulation or intubation) performed in the ICU may be a potential source of pain, therefore there is a clinical need for a simple and easy ICU pain scale to evaluate this condition in patients unable to self-report pain.

Assessment of pain in patients treated in the ICU becomes a daily clinical challenge for the ICU team, especially in those units where deep levels of sedation are used, but also in the minimal sedation environment based on analgesia. Various guidelines and recommendations exist to guide the ICU care team in the pain management and assessment process. Nevertheless, the gold standard for pain assessment is patient's self-report of pain (using numeric raing scale - NRS or visual analog scale - VAS), which can be aided with behavioural scales only when the self-report is unreliable or impossible to obtain. Those observational pain scales include the Critical-Care Pain Observation Tool (CPOT) and the Behavioural Pain Scale (BPS) and have been recommended for clinical use in the critically ill adults. However, their validation in a given patient population (cardiac, burn, different languages) is strongly recommended and required.

The need to equip critical care teams with dedicated monitoring tools is clear as early identification warrants early treatment. The CPOT has been developed by ICU professionals, yet it has not been translated or validated in Polish until now.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years,
* Ability to communicate in the Polish language,
* Intubated or with tracheostomy for more than 48 hours before inclusion with or without mechanical ventilation (controlled modes, spontaneous modes),
* Richmond Agitation Sedation Scale (RASS) above or equal to -3,
* Unrestricted sight and hearing,
* No limitations for body position changing,
* With no important intervention within last 48 hours prior to inclusion into the study (i.e. operation, tracheostomy).

Exclusion Criteria:

* A medical need for deep sedation - treatment of severe respiratory failure associated with patient-ventilator dyssynchrony, preventing awareness during neuromuscular blockade, status epilepticus, certain surgical conditions requiring immobility , cases of severe brain injury with intracranial hypertension
* Facial trauma (unable to evaluate facial expression),
* Richmond Agitation Sedation Scale (RASS) -4 or -5
* Neurological or psychiatric disorders,
* Use of neuromuscular blocking agents,
* Regular narcotic users,
* Chronic pain syndrome patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated adult ICU patients at the Intensive Care Unit of the Department of Anaesthesia, Intensive Care and Acute Poisoning of the tertiary teaching hospital at the Pomeranian Medical University in Szczecin, Poland undergoing minimal analgesia-based sedation protocol (fentanyl or morphine intravenous infusion).
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Interrater variability for Polish CPOT | Through study completion and up to 24 weeks.

SECONDARY OUTCOMES:
Criterion validity for Polish CPOT | Through study completion and up to 24 weeks.
Discriminant validity for Polish CPOT | Through study completion and up to 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna L Kotfis, MD,PhD, Principal Investigator — Pomeranian Medical University
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No